CLINICAL TRIAL: NCT07118618
Title: Probenecid, Pannexin 1 Channels for Alcohol Use Disorder
Brief Title: Probenecid Administration for Alcohol Craving and Consumption
Acronym: PROB2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Associate Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00000881
Record Dates: First submitted 2025-07-31; First posted 2025-08-12 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol Consumption; Craving
Keywords: AUD; Probenecid; Craving; Alcohol
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Probenecid

STUDY DESIGN:
Intervention Model Description: 16-week, between-subject, double-blind, randomized controlled trial (RCT) with probenecid (2g /day) compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug (Experimental): Probenecid 2gr oral
  Interventions: Drug: Probenecid Oral Tablet
- Placebo (Placebo Comparator): Placebo inactive
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Probenecid Oral Tablet — 2gr daily
  Other Names: Probalan
  Arms: Study drug
Drug: Placebo Oral Tablet — Inactive compound
  Other Names: Matching Inactive Oral Tablet
  Arms: Placebo

SUMMARY:
This study proposes a 16-week, between-subject, double-blind, randomized controlled trial (RCT) with probenecid (2g /day) compared to placebo in individuals with AUD to test if reduces craving and alcohol consumption.

DETAILED DESCRIPTION:
There are three aims in this study that test the hypothesis that probenecid compared to placebo, decreases:

* Aim 1 (laboratory phase): acute alcohol craving.
* Aim 2 (naturalistic phase): alcohol craving.
* Aim 3 (naturalistic phase): alcohol consumption

ELIGIBILITY:
Inclusion Criteria:

* • Male or female, ≥18 years.

  * women >7 drinks/week; men >14 drinks/week.
  * meet moderate to severe AUD score for DSM-5 criteria.
  * Breath Alcohol Content (BrAC)=0.00 at each visit.
  * in good health as confirmed by medical history, physical examination and lab tests.
  * willing to adhere to the study procedures.
  * understand informed consent and questionnaires in English at an 8th grade level.

Exclusion Criteria:

* • Women who are breastfeeding or positive urine test for pregnancy.

  * clinically significant medical abnormalities: unstable hypertension, clinically significant abnormal EKG, bilirubin >150% of the upper normal limit, ALT/AST >300% the UNL, creatinine clearance ≤60 dl/min
  * meet DSM-5 criteria for a diagnosis of schizophrenia, bipolar disorder, or other psychoses
  * medications that reduce alcohol consumption (naltrexone, disulfiram).
  * use aspirin (salicylates may reduce effect of probenecid), penicillin, methotrexate (may increase concentration).
  * history of suicide attempts in the last three years.
  * current diagnosis of a moderate or severe cannabis use disorder as assessed by self-report, SCID-E for SUD, and urine toxicology screen at baseline.
  * current diagnosis of another substance disorder at any severity, other than nicotine, as assessed by self-report, SCID-E for SUD, and urine toxicology screen at baseline.
  * current use of medications that may interact with probenecid.
  * history of hypersensitivity to sulfa drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Alcohol Craving | 5- week
  Acute alcohol craving during an alcohol cue-reactivity procedure assessed using change in the alcohol urge questionnaire (AUQ). AUQ consists of eight statements about the respondent's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). Drinking refers to various types of alcohol, including beer, wine and liquor. The respondent is asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "strongly disagree" to "strongly agree." Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Minimum score is 7, maximum score is 48. Higher scores reflect greater alcohol craving (worse outcome)

SECONDARY OUTCOMES:
Alcohol craving | 12-week
  Alcohol craving in naturalistic condition will be measured using craving the Obsessive Compulsive Drinking Scale (OCDS). The OCDS is a 14-item questionnaire, each rated on a scale from 0 to 4 that measures individuals' alcohol use and their attempts to control their drinking. Range Min score 0; max score. OCDS can also divided into two subscales: Obsessive subscale (items 1-6): max score = 24; Compulsive subscale (items 7-14): max score = 32. Higher scores reflect greater alcohol craving (worse outcome). Each item contributes equally to the total, and higher scores reflect greater obsessive and compulsive thoughts and behaviors related to alcohol use.

OTHER OUTCOMES:
Alcohol consumption | 12-week
  Number of standard drinks per week (DPW) in naturalistic condition as measured by the timeline follow-back (TLFB)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Haass-Koffler, PharmD, PhD, Principal Investigator — Brown Univiversity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hornbacher R, Gully BJ, Brown ZE, Brown JC, Magill M, Cioe PA, Swift RM, Sanna PP, Haass-Koffler CL. Probenecid as a pharmacotherapy for alcohol use disorder: A randomized placebo-controlled alcohol interaction trial. Alcohol Clin Exp Res (Hoboken). 2024 Dec;48(12):2391-2403. doi: 10.1111/acer.15470. Epub 2024 Oct 29. PMID 39472130